CLINICAL TRIAL: NCT05021783
Title: Investigation of the Relationship Between Sacroiliac Magnetic Resonance Imaging (MRI) Scores and Quantitative Sensory Testing in Patients With Axial Spondyloarthritis
Brief Title: The Relationship Between Magnetic Resonance Imaging (MRI) Scores and Sensory Testing in Axial Spondyloarthritis
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2021.64
Record Dates: First submitted 2021-08-16; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Central Sensitisation; Axial Spondyloarthritis; Inflammation
MeSH Terms: conditions — Axial Spondyloarthritis; Inflammation | interventions — Postsynaptic Potential Summation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with Axial SpondyloArthritis
  Interventions: Diagnostic Test: Pressure pain threshold; Diagnostic Test: Central Sensitization Inventory; Other: Spondyloarthritis Research Consortium of Canada scoring system; Diagnostic Test: Temporal Summation; Diagnostic Test: Conditioned pain modulation

INTERVENTIONS:
Diagnostic Test: Pressure pain threshold — The sacroiliac PPT scores will be obtained bilaterally from four measurement points; the first point is located 1 cm medially and caudally from spina iliaca posterior superior (SIPS) and 3 more laterally, medially and cranially.The left trapezius muscle will be used to evaluate distant control point .The 1 cm2 algometer probe will be placed vertically in the each selected point and pressure will be increased with 0.1 kg/sc until the participant reporting pressure became painful. The pressure value at which the pain is first felt will be accepted as the PPT of that point.
  Other Names: PPT
Diagnostic Test: Central Sensitization Inventory — Standardized questionnaire to determine the level of central sensitization
  Other Names: CSI
Other: Spondyloarthritis Research Consortium of Canada scoring system — SPARCC scoring consists of two subcomponents to detect sacroiliitis activation and structural damage. In the short tau inversion recovery (STIR) sequence, 6 consecutive coronal sections will be examined and the signal increase will be scored as 0 = normal signal and 1 = increased signal. In this way, the maximum score can be 12 in a single coronal section. Evaluations Total maximum score of 72 in 6 consecutive coronal sections. In structural scoring, similar to sacroiliitis scoring, the SI joint is divided into four quadrants to evaluate whether there is fatty change, erosion, backfill and ankylosis. Each lesion is scored as 0=absent or 1=present. In this way, fatty change and erosion can be scored between 0-40 and backfill and ankylosis can be scored between 0-20 in 5 consecutive sections in total scoring.
  Other Names: SPARCC
Diagnostic Test: Temporal Summation — TS will be evaluated over the trapezius muscle and sacroiliac joints with manuel algometer. In the evaluation of TS, a pressure as much the PPT value of each point will be applied with pain pressure algometer ten times with a 1-second interstimulus interval. Patients will be asked to rate their pain using on a 0 to 10 visual analogue scale (VAS) at 0, 5, and 10 seconds. TS will be calculated by subtracting the rating at 0 seconds from the rating at 10 seconds. The point that is located 1 cm medially and caudally from SIPS was used for SI joint TS measurement on both sides.
  Other Names: TS
Diagnostic Test: Conditioned pain modulation — First stimulus will be applied to trapezius with the pressure that induced a pain intensity of 4 point on a 10 point VAS as called a test stimulus. After that the right hand of the patient will be immersed in 7 Celsius water for 20 seconds to create a conditioning stimulus. Second test stimulus with the same intensity of first one will be applied to trapezius after the conditioning stimulus and patients will be asked to rate their pain. If the patients cannot hold their hand in the water for 20 seconds, the test stimulus will be applied immediately after the patients removed their hands out of water. The ratio between the first and second VAS values multiplied by 100 will be defined as CPM score
  Other Names: CPM

SUMMARY:
Axial spondyloarthritis is one of the most common rheumatic diseases and chronic pain and morning stiffness are the main complaints of these patients. Central sensitization is defined as increased response to normal or sub-threshold stimuli of central nervous system and its close relationship with many rheumatological diseases has been demonstrated in several studies. There is no method for the diagnosis of central sensitization is accepted as a gold standard. The clinical scales and quantitative sensory testing (QST) widely is used for this purpose widely. The most commonly used QST types include pressure pain threshold (PPT), temporal summation (TS) and conditioned pain modulation (CPM). The well-known scale used for the evaluation of central sensitization is the Central Sensitization Inventory (CSI) , developed in 2011 for detect central sensitization in chronic pain patients. In this study, it was aimed to investigate the relationship between QST and CSI and sacroiliac MRI changes.

DETAILED DESCRIPTION:
Central sensitization is hypersensitivity and increased response to normal/painless stimuli due to dysfunction in endogenous pain pathways. Quantitative sensory testing is frequently used to detect pain sensitization, and pressure pain threshold (PPT) and temporal summation (TS) are often preferred for this purpose. Recently, in addition to these methods, conditional pain modulation (CPM), in which descending pain pathways are tested, is also preferred. With PPT and TS measurement, local/generalized sensitivity increase can be detected in patients who develop pain sensitization. Observation of increased nociceptor response and decrease in pressure pain threshold in the tissue damaged area is interpreted in favor of peripheral sensitization, while obtaining a similar response in adjacent or distant areas is defined as generalized increased sensitivity. Although it is known that local hyperalgesia is one of the main findings of inflammation, studies that have shown this quantitatively are limited. Inflammatory lesions are observed in patients with axial spondyloarthritis, especially in the active stages of the disease, and the relationship of these lesions with PPT, TS and CPM values and pain sensitization is unknown. Therefore, in this study, it was planned to investigate the relationship of inflammatory and structural lesions detected by sacroiliac MRI with regional PPT,TS, CPM and pain sensitization in patients diagnosed with axSpA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with axSpA according to the Assessment of SpondyloArthritis International Society (ASAS) criteria
* Aged between 18-65 years

Exclusion Criteria:

* Had an other rheumatic diseases, peripheral vascular disease, peripheral neuropathy and spine disease (e.g., symptomatic herniated disc, spinal stenosis),
* Using centrally acting pain medications (e.g., pregabaline, duloxetine, opioids) or glucocorticoids (>10 mg prednisone or its equivalent) within 3 months of study enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AxSpA patientsThe patients aged 18-65 years diagnosed with axSpA according to the ASAS criteria will be recruited from a Rheumatology outpatient clinic of a single tertiary care hospital
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Central Sensitization Inventory (CSI) | 1 months
  25 somatic and psychosocial symptoms, which are frequently found in patients with central sensitization in part A, are questioned. In part B, the presence of diseases whose relationship with central sensitization is well defined is questioned in the patient without participating in scoring. Central sensitization is assumed in patients who score 40 or more over 100 points. As the score increases, the severity of sensitization is considered to increase.
Pressure pain threshold (PPT) | 1 months
  The sacroiliac PPT scores were obtained from four measurement points; the first point was located 1 cm medially and caudally from spina iliaca posterior superior (SIPS) and 3 more laterally, medially, and cranially. Lower scores are interpreted in favor of increased pain sensitization.
Temporal summation (TS) | 1 months
  TS will be evaluated over the trapezius muscle and sacroiliac joints with manuel algometer. In the evaluation of TS, a pressure as much the PPT value of each point will be applied with pain pressure algometer ten times with a 1-second interstimulus interval. Patients will be asked to rate their pain using on a 0 to 10 visual analogue scale (VAS) at 0, 5, and 10 seconds. TS will be calculated by subtracting the rating at 0 seconds from the rating at 10 seconds. The point that is located 1 cm medially and caudally from SIPS was used for SI joint TS measurement on both sides. As the score increases, the severity of sensitization is considered to increase.
Conditioned pain modulation (CPM) | 1 months
  First stimulus will be applied to trapezius with the pressure that induced a pain intensity of 4 point on a 10 point VAS as called a test stimulus. After that the right hand of the patient will be immersed in 7 Celsius water for 20 seconds to create a conditioning stimulus. Second test stimulus with the same intensity of first one will be applied to trapezius after the conditioning stimulus and patients will be asked to rate their pain. If the patients cannot hold their hand in the water for 20 seconds, the test stimulus will be applied immediately after the patients removed their hands out of water. The ratio between the first and second VAS values multiplied by 100 will be defined as CPM score. Higher scores indicate better descending pain inhibition.

SECONDARY OUTCOMES:
Spondyloarthritis Research Consortium of Canada (SPARCC) scoring system | 1 months
  SPARCC scoring consists of two subcomponents to detect sacroiliitis activation and structural damage.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kiltz U, Baraliakos X, Regel A, Buhring B, Braun J. Causes of pain in patients with axial spondyloarthritis. Clin Exp Rheumatol. 2017 Sep-Oct;35 Suppl 107(5):102-107. Epub 2017 Sep 29. PMID 28967358
- [Result] Classification of chronic pain. Descriptions of chronic pain syndromes and definitions of pain terms. Prepared by the International Association for the Study of Pain, Subcommittee on Taxonomy. Pain Suppl. 1986;3:S1-226. No abstract available. PMID 3461421
- [Result] Rolke R, Baron R, Maier C, Tolle TR, Treede -DR, Beyer A, Binder A, Birbaumer N, Birklein F, Botefur IC, Braune S, Flor H, Huge V, Klug R, Landwehrmeyer GB, Magerl W, Maihofner C, Rolko C, Schaub C, Scherens A, Sprenger T, Valet M, Wasserka B. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain. 2006 Aug;123(3):231-243. doi: 10.1016/j.pain.2006.01.041. Epub 2006 May 11. PMID 16697110
- [Result] Maksymowych WP, Inman RD, Salonen D, Dhillon SS, Williams M, Stone M, Conner-Spady B, Palsat J, Lambert RG. Spondyloarthritis research Consortium of Canada magnetic resonance imaging index for assessment of sacroiliac joint inflammation in ankylosing spondylitis. Arthritis Rheum. 2005 Oct 15;53(5):703-9. doi: 10.1002/art.21445. PMID 16208659
- [Result] Maksymowych WP, Wichuk S, Chiowchanwisawakit P, Lambert RG, Pedersen SJ. Development and preliminary validation of the spondyloarthritis research consortium of Canada magnetic resonance imaging sacroiliac joint structural score. J Rheumatol. 2015 Jan;42(1):79-86. doi: 10.3899/jrheum.140519. Epub 2014 Oct 15. PMID 25320219
- [Result] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Result] van Leeuwen RJ, Szadek K, de Vet H, Zuurmond W, Perez R. Pain Pressure Threshold in the Region of the Sacroiliac Joint in Patients Diagnosed with Sacroiliac Joint Pain. Pain Physician. 2016 Mar;19(3):147-54. PMID 27008288
- [Result] de Goeij M, van Eijk LT, Vanelderen P, Wilder-Smith OH, Vissers KC, van der Hoeven JG, Kox M, Scheffer GJ, Pickkers P. Systemic inflammation decreases pain threshold in humans in vivo. PLoS One. 2013 Dec 17;8(12):e84159. doi: 10.1371/journal.pone.0084159. eCollection 2013. PMID 24358337